CLINICAL TRIAL: NCT00392704
Title: A Phase II Trial of Neoadjuvant Chemotherapy Plus Bevacizumab Followed By Concurrent Chemotherapy/Bevacizumab/Erlotinib/Radiation Therapy in the Treatment of Locally Advanced Squamous Carcinoma of the Head and Neck
Brief Title: Treatment of Head & Neck Cancer With Chemotherapy and Radiation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI HN 08
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride; Paclitaxel; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): All patients initially received treatment with paclitaxel 200 mg/m2, 3 hour IV infusion days 1 and 22; carboplatin area under the curve (AUC) 6.0 IV, days 1 and 22; 5-fluorouracil (5-FU) 200 mg/m2 daily by 24-hour continuous IV infusion, days 1 to 43; bevacizumab 15 mg/kg IV infusion days 1 and 22.
  One to three weeks after completing neoadjuvant therapy, patients began treatment with concurrent chemoradiation, bevacizumab, and erlotinib. Radiation therapy began on day 1, with 1.8-Gy single daily doses, Monday through Friday, to a total dose of 68.4 Gy. Paclitaxel 50 mg/m2 was administered by 1-hour IV infusion on days 1 and 22. Erlotinib 150 mg by mouth daily began concurrently with radiation therapy and continued daily during the 7-week course of radiation.
  Interventions: Drug: Bevacizumab; Drug: Erlotinib; Drug: Paclitaxel; Drug: 5-FU; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Bevacizumab — Induction Treatment:
  Paclitaxel 200mg/m2 by vein over 1-3 hours on Day 1 & Day 22 Carboplatin AUC 6.0 by vein over 1 hour on Days 1 and 22 Bevacizumab 15mg/kg by vein over 60-90 minutes on Days 1 and 22 5-FU 200mg/m2 as a 24 hour continuous infusion via pump on Days 1 through 43.
  Combined Modality Treatment:
  Radiation therapy is given daily, Monday through Friday for approximately 7 weeks. Erlotinib 150mg by mouth daily during the entire course of radiation (approximately 7 weeks) Paclitaxel 50mg/m2 by vein over 1-hour weekly for 6 weeks beginning Day 1 of radiation therapy Bevacizumab 15mg/kg by vein over 30-90 minutes on Days 50 and 71 at the same time of radiation therapy
  Other Names: Avastin
Drug: Erlotinib — Induction Treatment:
  Paclitaxel 200mg/m2 by vein over 1-3 hours on Day 1 & Day 22 Carboplatin AUC 6.0 by vein over 1 hour on Days 1 and 22 Bevacizumab 15mg/kg by vein over 60-90 minutes on Days 1 and 22 5-FU 200mg/m2 as a 24 hour continuous infusion via pump on Days 1 through 43.
  Combined Modality Treatment:
  Radiation therapy is given daily, Monday through Friday for approximately 7 weeks. Erlotinib 150mg by mouth daily during the entire course of radiation (approximately 7 weeks) Paclitaxel 50mg/m2 by vein over 1-hour weekly for 6 weeks beginning Day 1 of radiation therapy Bevacizumab 15mg/kg by vein over 30-90 minutes on Days 50 and 71 at the same time of radiation therapy
  Other Names: Tarceva
Drug: Paclitaxel — Neoadjuvant: 200 mg/m2 IV, 1-3 hour infusion, Days 1 and 22
  Combined Modality: 50 mg/m2 IV, 1 hour IV infusion, weekly x6, beginning day 1 of radiation therapy
  Other Names: Taxol
Drug: 5-FU — Neoadjuvant: 200 mg/m2 24 hour continuous infusion days 1-43
  Other Names: 5-fluorouracil; Efudex
Radiation: Radiation Therapy — Combined Modality Therapy: 1.8 Gy/day, Monday-Friday, total dose 68.4 Gy
  Other Names: RT

SUMMARY:
Two new cancer treatment drugs called targeted therapies will be added to standard treatment for head and neck cancer to see if an improvement can be made in the effectiveness of treatment for this type of cancer. Treatment will include chemotherapy, radiation therapy and targeted therapy taken over a period of 4 months.

DETAILED DESCRIPTION:
In this trial, patients will receive induction treatment with combination chemotherapy(paclitaxel/carboplatin/infusional 5FU) plus bevacizumab. After 6 weeks of treatment, patients will be reevaluated and will then receive concurrent radiation therapy, chemotherapy (weekly paclitaxel),bevacizumab, and erlotinib.

Induction Treatment:

Paclitaxel 200mg/m2 by vein over 1-3 hours on Day 1 & Day 22 Carboplatin AUC 6.0 by vein over 1 hour on Days 1 and 22 Bevacizumab 15mg/kg by vein over 60-90 minutes on Days 1 and 22 5-FU 200mg/m2 as a 24 hour continuous infusion via pump on Days 1 through 43.

Combined Modality Treatment:

Radiation therapy is given daily, Monday through Friday for approximately 7 weeks. Erlotinib 150mg by mouth daily during the entire course of radiation (approximately 7 weeks) Paclitaxel 50mg/m2 by vein over 1-hour weekly for 6 weeks beginning Day 1 of radiation therapy Bevacizumab 15mg/kg by vein over 30-90 minutes on Days 50 and 71 at the same time of radiation therapy

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed head & neck cancer
* Considered low cure rate with local therapy
* No prior treatment for this cancer
* Able to be up & about and perform self care
* Adequate renal and liver function
* Must be 18 years of age or older
* All patients will need an indwelling central venous access catheter
* Must be able to give written informed consent

Exclusion Criteria:

* Active cancer treatment in the last 5 years
* Pregnant or lactating women
* History of stroke, transient ischemic attacks, or acute myocardial infarction within the past 6 months or any other serious cardiovascular disease
* History of neurological disease
* Recent history of blood in the sputum or vomitus
* Non-healing wounds, ulcer or long bone fractures
* History of bleeding problems or coagulation problems
* History of abdominal fistula, gastrointestinal perforation or intrabdominal abscess within 6 months
* History of uncontrolled hypertension
* Symptomatic peripheral vascular disease

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Background] Hainsworth JD, Spigel DR, Greco FA, Shipley DL, Peyton J, Rubin M, Stipanov M, Meluch A. Combined modality treatment with chemotherapy, radiation therapy, bevacizumab, and erlotinib in patients with locally advanced squamous carcinoma of the head and neck: a phase II trial of the Sarah Cannon oncology research consortium. Cancer J. 2011 Sep-Oct;17(5):267-72. doi: 10.1097/PPO.0b013e3182329791. PMID 21952273

RESULTS

PARTICIPANT FLOW:
Period: Neoadjuvant Chemotherapy
Arm/Group | Intervention
Started | 60
Completed | 54
Not Completed | 6
Period: Combined Modality Therapy
Arm/Group | Intervention
Started | 54
Completed | 49
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 60
Age Continuous [Median (Full Range); unit: years] | 56 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 50
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Two-Year Progression Free Survival (PFS) Probability, the Percentage of Patients Estimated to be Alive Without Worsening of Their Disease Two Years After Beginning Protocol Treatment
Description: The percentage of patients estimated to be alive 2 years after beginning protocol treatment
Time Frame: 24 months
Population: All participants in this study were assessed and included in the progression free survival analysis
Measure: Number; unit: percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 60
percentage of participants | 83

2. Secondary Outcome: Overall Survival (OS)Probability, the Percentage of Patients Estimated to be Alive Two Years After Beginning Protocol Treatment
Description: The Percentage of Patients Estimated to be Alive Two Years After Beginning Protocol Treatment
Time Frame: 24 Months
Measure: Number; unit: percentage of patients
Arm/Group | Intervention
Number analyzed (Participants) | 60
percentage of patients | 90

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 24/60
Other Adverse Events (participants affected / at risk) | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=60)
Leukocytes (Blood and lymphatic system disorders) | 1 (1)
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Weakness (General disorders) | 2 (3)
Diverticulitis (Gastrointestinal disorders) | 1 (2)
Pneumatosis Intestinalis (Gastrointestinal disorders) | 1 (1)
Mucositis/Stomatitis (Gastrointestinal disorders) | 4 (5)
Dehydration (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fistula, GI (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 3 (3)
Infection - Sepsis (Infections and infestations) | 1 (1)
Infection with Unknown ANC (Infections and infestations) | 2 (2)
Hemorrhage with Surgery (Surgical and medical procedures) | 1 (2)
Infection - Pneumonia (Infections and infestations) | 2 (2)
CNS Ischemia (Vascular disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=60)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 32 (67)
ALT (Metabolism and nutrition disorders) | 5 (7)
Anorexia (Gastrointestinal disorders) | 33 (52)
AST (Metabolism and nutrition disorders) | 8 (8)
Bilirubin (Metabolism and nutrition disorders) | 6 (6)
Rigor/Chills (General disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 25 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Creatinine (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 38 (55)
Dermatitis (Skin and subcutaneous tissue disorders) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 38 (69)
Dizziness (Nervous system disorders) | 9 (15)
Dry Mouth (Gastrointestinal disorders) | 13 (17)
Dry Skin (Skin and subcutaneous tissue disorders) | 9 (12)
Dysphagia (Gastrointestinal disorders) | 25 (30)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Edema - Neck (Blood and lymphatic system disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 12 (18)
Esophagitis (Gastrointestinal disorders) | 15 (17)
Fatigue (General disorders) | 44 (105)
Fever (General disorders) | 17 (22)
Hand-Foot Syndrome (Skin and subcutaneous tissue disorders) | 13 (20)
Hemoglobin (Blood and lymphatic system disorders) | 39 (72)
Hemorrhage - Nose (Blood and lymphatic system disorders) | 11 (14)
Hemorrhoids (Gastrointestinal disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Cardiac disorders) | 5 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (6)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6)
Hypotension (Cardiac disorders) | 7 (8)
Infection - NOS (Infections and infestations) | 6 (6)
Infection - PEG Site (Infections and infestations) | 8 (9)
Infection - Throat (Infections and infestations) | 6 (10)
Insomnia (General disorders) | 14 (21)
Leukocytes (Blood and lymphatic system disorders) | 40 (81)
Malnutrition (Metabolism and nutrition disorders) | 3 (4)
Mood Alteration - Anxiety (Psychiatric disorders) | 8 (16)
Mood Alteration - Depression (Psychiatric disorders) | 7 (11)
Mucositis/Stomatitis (Gastrointestinal disorders) | 57 (118)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 37 (65)
Neutrophils (Blood and lymphatic system disorders) | 43 (60)
Pain - NOS (General disorders) | 51 (127)
Pain - Joint (General disorders) | 3 (4)
Platelets (Blood and lymphatic system disorders) | 27 (46)
Proteinuria (Metabolism and nutrition disorders) | 8 (12)
Pruritis (Skin and subcutaneous tissue disorders) | 8 (8)
Burn (Skin and subcutaneous tissue disorders) | 11 (13)
Acne (Skin and subcutaneous tissue disorders) | 4 (4)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 44 (89)
Reflux (Gastrointestinal disorders) | 4 (6)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Neuropathy - Sensory (Nervous system disorders) | 26 (48)
Superventricular Arrhythmia (Cardiac disorders) | 4 (5)
Sweating (General disorders) | 3 (3)
Syncope (Nervous system disorders) | 3 (3)
Taste Alteration (Gastrointestinal disorders) | 16 (22)
Vomiting (Gastrointestinal disorders) | 25 (33)
Weight Loss (Metabolism and nutrition disorders) | 25 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.